CLINICAL TRIAL: NCT02548507
Title: Prevalence, Main Features and Treatment of Nocturnal Leg Cramps in Geneva: A Primary Care Prospective Observational Study
Brief Title: Nocturnal Leg Cramps in Geneva : an Observational Study
Acronym: CNMI
Status: Completed | Type: Observational
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Maisonneuve Hubert, Maitre d'enseignement et de recherche, University of Geneva, Switzerland
Other Study IDs: CNMI
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Sleep Wake Transition Disorders; Nocturnal Leg Cramps
MeSH Terms: conditions — Sleep-Wake Transition Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational study, no intervention

SUMMARY:
Background :

Nocturnal leg cramps (NLC) are defined as painful involuntary contractions of the lower limbs occurring during prolonged periods of rest, typically during the night. They may cause severe pain and sleep disturbance, and are particularly common among older adults, though they can occur in all decades of life. They are frequently unreported to physicians. To the investigators' knowledge, no epidemiological studies have been conducted in Switzerland, but in a general population survey carried out in the UK (n=233), the overall prevalence of NLC was 37% and the disorder was more prevalent in older subjects (>80 years old: 54%). Of those who experienced NLC, 40% had cramps three or more times per week and 6% nightly. Another study performed in older US veterans (n=515) showed that 56% suffered from NLC.

The precise cause of these cramps is unclear. Most NLC occurring in adults appear to be idiopathic, but potential contributing factors include low levels of certain minerals, extracellular fluid volume depletion and prolonged sitting or inappropriate leg position during sedentary activity.

Research question :

What are the prevalence and the main features of NLC in patients consulting primary care physicians (PCPs) in Geneva, and how do PCPs treat this affection?

Primary objective :

To compute the prevalence of NLC in patients consulting PCPs in Geneva, explore its main features (number, duration, severity and sleep disturbance) and assess how PCPs treat this affection.

Study design :

Prospective observational study using questionnaire and daily log completed by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 50 years old or more,
* currently presenting NLC (The definition of NLC used for the purpose of the study is any cramp in the legs or feet, occurring during the sleep (eg long rest) period).
* coming to the practice for a planned consultation.

Exclusion Criteria:

* Patients suffering from a terminal illness
* from disorders affecting their ability to consent,
* not speaking French
* or not having a telephone.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 50 years old or more, consulting primary care physicians in Geneva
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of NLC | Presence or absence of NLC will be checked during the time of recruitment for each participant PCP, with expected average of 1 to 6 months.
  In order to compute the prevalence of NLC, the PCPs will be asked to specify for each patient coming for a planned consultation whether he/she has NLC, meets the inclusion criteria and accept to participate (group 1), has NLC, meets the inclusion criteria but refuses to participate (group 2) or has NLC but does not meet the inclusion criteria (group 3). For patients in the group 1 doctors will record the current date, the name and the first name, the gender, the date of birth and the phone number; for patients in the group 2 they will record the current date, the gender and the date of birth; and finally for patients in the group 3 they will record the current date, the gender, the date of birth and the exclusion criterion.

SECONDARY OUTCOMES:
Frequency of NLC | During two weeks after recruitment
  Voluntaries will record during two weeks the number of cramps in a daily log.
Duration of nocturnal leg cramps | During two weeks after recruitment
  Voluntaries will record during two weeks the duration of cramps in a daily log.
Severity of pain related with nocturnal leg cramps | During two weeks after recruitment
  Voluntaries will record the severity of cramps in a daily log, standardized on an analog numerical scale of 1 to 10 .
Severity of sleep disturbance related with nocturnal leg cramps | During two weeks after recruitment
  Voluntaries will record the severity of sleep disturbance related with NLC, in a daily log, standardized on an analog numerical scale of 1 to 10.
Patient expectancies for nocturnal leg cramps treatment | Two weeks after recruitment
  We will ask the voluntaries to specify the average pain and sleep disturbance related with NLC on analog numerical scale of 1 to 10. We'll then ask them what improvement they would expect from a treatment on the same analog numeric scale for pain and sleep disturbance.
Patient quality of life | 1 year after initial recruitment
  Voluntaries will fill a SF36 questionnaire
Patient quality of sleep | 1 year after initial recruitment
  Voluntaries will fill a PSQI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Maisonneuve, MD, Principal Investigator — University of Geneva
Locations (1):
- Primary care network, Geneva, Switzerland